CLINICAL TRIAL: NCT03541148
Title: Evaluation of the Nutritional Supplement Oncoxin-Viusid® in the Treatment of 20 Patients With Cutaneous Melanoma in Stage IIB-IIIA
Brief Title: Evaluation of Oncoxin-Viusid® in Cutaneous Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-2
Record Dates: First submitted 2018-05-03; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Cutaneous Melanoma, Stage II; Malignant Cutaneous Melanoma; Cutaneous Melanoma, Stage III
Keywords: Cutaneous malignant melanoma; Nutritional supplement; survival; Green tea
MeSH Terms: conditions — Melanoma; Melanoma, Cutaneous Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncoxin-Viusid (Experimental): Nutritional supplement Oncoxin-Viusid 25 mL in oral solution twice a day
  Interventions: Dietary Supplement: Oncoxin-Viusid

INTERVENTIONS:
Dietary Supplement: Oncoxin-Viusid — Oncoxin-Viusid supplement before/during/after standard surgical and adjuvant treatment or chemotherapy.

SUMMARY:
Malignant melanoma, responsible for 75% of deaths from skin cancer. Current therapeutic options have poor response, many adverse events and high costs. For this reason, a study with nutritional supplement Oncoxin-Viusid was carried out. According to previous studies, it has an antitumor, immunomodulatory effect and to potentiate the antiproliferative effect of standard chemotherapeutic agents in different locations and stages of cancer.

DETAILED DESCRIPTION:
Performed at Manuel Fajardo Surgical Clinical University Hospital in Havana, Cuba from September 2014 to April 2018, following a proof of concept open label study, with no control group in 20 patients diagnosed histologically in Fajardo Hospital or Oncology Institute, as Melanoma, primary cutaneous stage IIB-IIIA. All received conventional surgical treatment and oral Oncoxin-Viusid (25 ml 2 times a day for one year), where it was also indicated adjuvant treatment or chemotherapy. All were evaluated monthly the first year and semesterly the second year. Complying with the provisions of the Helsinki Act.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of Malignant Cutaneous Melanoma in stage IIB-IIC-IIIA
* Subjects of 18 years and over of both sexes.
* General health status according to the Karnofsky Index ≥ 70.
* Laboratory parameters within the normal limits defined as: Hematopoietic: Hemoglobin ≥ 9 g / L, Total Leukocytes ≥ 3 x 109 cells / L, Neutrophils ≥ 1.5 x 109 cells / L, Platelets ≥ 100 x 109 / L Hepatic: Liver function within 2.5 times upper normal limit and without liver disease demonstrated by TGP, OGT and alkaline phosphatase.
* Patients who express written voluntariness to enter the study with their signature of the informed consent document.
* Women of childbearing age should have a negative pregnancy test and use effective contraceptive methods such as intrauterine devices, hormonal contraceptives, barrier method or tubal ligation.

Exclusion Criteria:

* Pregnancy or lactation.
* Patients with a second concomitant tumor.
* Present an associated chronic disease in the decompensation phase (heart disease, diabetes, hypertension).
* History of hypersensitivity to another similar product.
* Severe acute allergic states.
* Severe septic processes.
* Non-operated patients, in whom the surgery was contraindicated.
* Patients at potential risk of not completing the study (those who will travel during the period of the investigation or distance in their residence, outside the city).
* Subjects who are participating in another clinical trial.
* Patients with cognitive disorders or a mental disorder that hinders their follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 2 years
  Calculated according to the method of Kaplan Meyer
Disease free survival rate | 2 years
  Calculated according to the Kaplan Meyer method

SECONDARY OUTCOMES:
Temporary interruption of conventional treatment | 2 years
  Due to adverse events
Presence of adverse events | 2 years
  Associated with conventional treatment
Type of adverse events | 2 years
  According to severity and causality
Quality of life | 2 years
  Quality of life questionnaire of the EORTC: QLQ30

CONTACTS AND LOCATIONS:
Overall Officials: Olaine R. Gray Lovio, Dr., Principal Investigator — Manuel Fajardo Clinical Surgical University Hospital
Locations (1):
- Manuel Fajardo Clinical Surgical University Hospital, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR